CLINICAL TRIAL: NCT00871195
Title: Evaluation Of The Performance Of A Noninvasive Test For Fetal RHD Genotype On The Sequenom MassARRAY System
Brief Title: A Noninvasive Test for Fetal RHD Genotype
Acronym: NAFTnet RHD
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Collaborators: NAFTNet (Other)
Responsible Party: Sponsor
Other Study IDs: SQNM-RHD-301
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Rhesus D Genotype
Keywords: Rhesus D; RHD; genotype; phenotype; neonatal; noninvasive; fetal; MassARRAY; DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat.
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to evaluate the performance of Sequenom's noninvasive test for fetal RHD genotype. The test uses MALDI-TOF mass spectrometry to detect DNA. The study is specifically designed to determine whether RHD typing using free fetal DNA in maternal circulation can accurately predict the neonatal RhD phenotype at birth.

DETAILED DESCRIPTION:
In the United States and Canada, routine obstetrical care includes a blood test to determine the blood type of the mother (ABO and RhD). An antibody screen for anti-red cell antibodies in the mother's serum is also performed.

Postpartum prophylactic treatment of RhD negative women with anti-D immunoglobulin to prevent "RhD Disease", or hemolytic disease of the fetus/newborn, was initiated in the 1960's. In the mid 1980's, the routine administration of antenatal anti-D immunoglobulin became the standard of care as well. Although these treatments have dramatically reduced the incidence of RhD Disease, approximately 40% of all RhD negative pregnancies continue to receive unnecessary injections of antenatal anti-D immunoglobulin.

Genotyping platforms such as MALDI-TOF mass spectrometry allow for precise and sensitive detection of fetal-specific (paternally derived) alleles in maternal plasma. In this study, Sequenom's MassARRAY technology will be used to assess a noninvasive test for fetal RHD genotyping in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Female at least 18 years of age
* RhD negative by serology
* Pregnant at no more than 11-13 weeks gestation confirmed by ultrasound
* Willing to provide signed and dated informed consent
* Able and willing to comply with the protocol

Exclusion Criteria:

* RhD negative women known to be alloimmunized to the RhD antigen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women who are known to be serologically RhD negative.
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To test as to whether advancing gestational age is associated with accuracy of fetal typing for RhD. | First, second, and third trimester

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Moise, MD, Principal Investigator — Baylor College of Medicine
Locations (13):
- United States (10):
  - Obstetrix Medical Group of Phoenix, Phoenix, Arizona
  - Wayne State University, Detroit, Michigan
  - Mt. Sinai School of Medicine, New York, New York
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Evergreen Hospital, Kirkland, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - Mt. Sinai School of Medicine, Toronto, Ontario
  - McGill University, Montreal, Quebec